CLINICAL TRIAL: NCT00508768
Title: A Randomized, Double-Blind, Parallel-Group, Pharmacokinetic Study of Oral SCIO-469 (90 mg qd and 30 mg Tid) in Female Subjects With Active Rheumatoid Arthritis
Brief Title: A Study of Oral SCIO-469 Pharmacokinetics (Study of a Drug in the Body to Watch How the Drug is Absorbed, Distributed, Metabolized and Eliminated Over a Period of Time) in the Body of Female Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005155
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — SCIO-469

INTERVENTIONS:
Drug: Oral SCIO-469 capsule

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of two oral dosing regimens of SCIO-469, with and without methotrexate, in patients with active rheumatoid arthritis.

DETAILED DESCRIPTION:
SCIO-469 is being developed for the treatment of active rheumatoid arthritis, a disease that occurs mostly in women; therefore, female patients with active rheumatoid arthritis are selected as the study population. This study is the first detailed pharmacokinetic evaluation (study of a drug in the body to watch how the drug is absorbed, distributed, metabolized and eliminated over a period of time) of SCIO-469 in a new capsule formulation. Methotrexate is frequently prescribed as treatment for patients with rheumatoid arthritis; thus, SCIO-469 could potentially be used along with methotrexate. It is not known how methotrexate affects the pharmacokinetics of SCIO-469; therefore, the study is designed to include patients who are taking stable doses of methotrexate and patients who are not taking methotrexate. This is a Phase II, randomized (study medication assigned by chance), double-blind (neither the patient or the physician knows which study treatment the patient is receiving), parallel-group study designed to assess the pharmacokinetics, safety, and tolerability of SCIO-469 in female patients with active rheumatoid arthritis. Sixteen patients will be enrolled in the study, with eight receiving stable doses of methotrexate and eight not receiving methotrexate. No other disease-modifying anti-rheumatic drugs (DMARDs) are allowed. Pharmacokinetics will be evaluated for SCIO-469 and its metabolites, testing for significant differences by occasion (Day 1 or Day 12), treatment (30 mg three times a day or 90 mg once a day), and stratum (methotrexate or non methotrexate). Safety assessments for this study include clinical adverse events, concomitant medications, and clinical assessments (medical history, physical examination, vital and orthostatic vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory evaluations [serum chemistry, urinalysis, hematology, liver function and other tests, and pregnancy test]). Patients receiving stable doses of methotrexate (taken once a week, either orally or by injection) and those not receiving methotrexate will be randomized into one of two oral capsule SCIO-469 dosing regimens: 30 mg three times a day and 90 mg once a day. Patients will take study drug for 11 of 12 days, with no study drug taken on Day 2. On Day 19, seven days after the end of treatment, patients will undergo a follow-up assessment of safety variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active rheumatoid arthritis
* Patients on methotrexate are required to have taken a stable methotrexate dose of 15 to 25 mg/week (or lower maximum-tolerated dose level) for at least 1 month before study entry
* Patients with no methotrexate are required to have taken no methotrexate for at least 1 month before study entry
* Non steroidal anti inflammatory drugs (NSAIDs) and low-dose prednisone are allowed if doses had been stable for at least 1 month before study entry
* Patients of childbearing potential must have agreed to practice two forms of birth control for the duration of the trial.

Exclusion Criteria:

* Have taken infliximab or experimental biological antagonists (e.g., TNF antagonists) within the 3-month period before study entry
* Have used leflunomide within the 3 month period before study entry
* Have taken etanercept, anakinra, and disease-modifying anti-rheumatic drugs (DMARDs) other than leflunomide (and methotrexate) within the 4-week period before study entry
* Received intra-articular, intramuscular, or intravenous (IV) doses of corticosteroids or received oral doses of corticosteroids exceeding 10 mg/day within the 4-week period before study entry
* Elevated levels (greater than 1.2 times the upper limit of normal) of aspartate transaminase or alanine transaminase within the 6-month period before study entry.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters will be evaluated for SCIO-469 and its metabolites, testing for significant differences by occasion (Day 1 or Day 12), treatment (30 mg three times a day or 90 mg once a day), and stratum (methotrexate or non methotrexate).

SECONDARY OUTCOMES:
Safety variables will be assessed on Day 19, seven days after the end of treatment, and will include adverse events, concomitant medications, and clinical assessments (medical history, physical exam, vital signs, 12-lead ECG, and clinical labs).

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.

REFERENCES:
- See also: A Pharmacokinetic Study of Oral SCIO-469 in Female Subjects with Active Rheumatoid Arthritis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=957&filename=CR005155_CSR.pdf